CLINICAL TRIAL: NCT01576029
Title: Phase II Randomized Study of Continuing Treatment With Docetaxel Versus Switching to Cabazitaxel After Minor Prostate Specific Antigen Response to Docetaxel in the First Line Treatment of Patients With Castration-Resistant Metastatic Prostate Cancer.
Brief Title: Continued Treatment With Docetaxel Versus Switch to Cabazitaxel After Minor Prostate Specific Antigen Response to Docetaxel in Patients With Castration-Resistant Metastatic Prostate Cancer
Acronym: SWITCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABAZ_L_05933; U1111-1119-8381 (Other: UTN)
Record Dates: First submitted 2012-03-30; First posted 2012-04-12 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel (Active Comparator): 75 mg/m2, administered as a 1-hour intravenous infusion, every 3 weeks
  Interventions: Drug: DOCETAXEL (XRP6976)
- Cabazitaxel (Experimental): 25 mg/m2, administered as a 1-hour intravenous infusion, every 3 weeks
  Interventions: Drug: CABAZITAXEL (XRP6258)

INTERVENTIONS:
Drug: CABAZITAXEL (XRP6258) — Pharmaceutical form: solution Route of administration: intravenous
  Arms: Cabazitaxel
Drug: DOCETAXEL (XRP6976) — Pharmaceutical form: solution Route of administration: intravenous
  Arms: Docetaxel

SUMMARY:
Primary Objective:

* To compare the continuation of treatment with docetaxel versus switching to cabazitaxel regarding the time to PSA (Prostatic Specific Antigen) progression (TTP-PSA), in patients with Castration-Resistant Prostate Cancer (CRPC) that, after four cycles of docetaxel, have minor PSA response (defined as a reduction between 1% and 49%) or increase of up to 24% in PSA levels.

Secondary Objectives:

* PSA response rate
* Overall survival (OS)
* Incidence of Adverse Events

DETAILED DESCRIPTION:
Screening: 21days (+7 days) Treatment: until PSA progression Post-treatment Follow-up: 2 years

ELIGIBILITY:
Inclusion criteria :

* Documentation of histological prostate cancer;
* Patients with metastatic CRPC (Castration-Resistant Metastatic Prostate Cancer) who progressed with hormone deprivation, including the withdrawal of antiandrogen-class drugs for at least 4 weeks, and 6 weeks for bicalutamide or if documented that PSA did not decrease during 3 months of this therapy;
* Documentation of metastasis by imaging (computerized tomography [CT], magnetic resonance imaging [MRI] or bone scan), in patients with PSA < 20 ng/mL at the time of inclusion
* Provide minor PSA response (characterized by a reduction between 1% and 49%) or increase up to 24% in PSA levels, in relation to the value measured before starting docetaxel therapy, measured at least 7 days after the fourth cycle of docetaxel;
* Patient has received 4 cycles of docetaxel at a dose of 75 mg/m2 ;
* ECOG performance status of 0 or 1;
* Marrow, liver and renal function within acceptable values;
* PSA ≥ 2 ng/mL;
* Testosterone level ≤ 50 ng/dL (for patients with no prior history of orchiectomy).

Exclusion criteria:

* Prior use of chemotherapy, except for docetaxel for four cycles;
* Documented disease progression during treatment with docetaxel (first 4 cycles);
* Patients with metastases resulting in neurological damage;
* Inability to continue receiving gonadotropin-releasing hormone agonists in patients with no prior history of orchiectomy;
* Use of recombinant methionyl human granulocyte-colony stimulating factor non-glycosylated (G-CSF) in the 24 hours preceding baseline;
* Any other current neoplasia or over the past 5 years, except for basal cell skin carcinoma or squamous skin cell carcinoma;
* Known seropositivity for HIV (Human immunodeficiency Virus );
* Concomitant diseases, such as significant neurological or psychiatric disease; uncontrolled hypercalcemia or any other serious comorbidity;
* Hypersensitivity or allergy to any of the study treatments.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Median time to PSA progression | up to 60 days

SECONDARY OUTCOMES:
PSA response rate: Percentage of patients with a decrease of at least 50% in the PSA | up to 60 days
Overall Survival: Median time elapsed between the date of starting treatment until death by any cause | up to a maximum of 2 years
Number of patients with adverse events | up to a maximum of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Brazil (8):
  - Investigational Site Number 004, Barretos
  - Investigational Site Number 008, Brasília
  - Investigational Site Number 009, Londrina
  - Investigational Site Number 003, Mogi das Cruzes
  - Investigational Site Number 005, Porto Alegre
  - Investigational Site Number 006, Rio de Janeiro
  - Investigational Site Number 001, Rio de Janeiro
  - Investigational Site Number 007, São Paulo